CLINICAL TRIAL: NCT03583658
Title: A Randomised, Double-blind, Placebo Controlled, Parallel Group, Multicentre Trial to Assess the Efficacy and Safety of Ambroxol Lozenges 20 mg (Hard Boiled Lozenges) Versus Placebo for the Relief of Sore Throat Pain in Patients With Acute Pharyngitis
Brief Title: Efficacy and Safety Study of New Ambroxol Hardboiled Lozenges in Acute Pharyngitis
Acronym: DELICIOUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPS15328; U1111-1202-9392 (Other: UTN)
Record Dates: First submitted 2018-06-18; First posted 2018-07-11 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ambroxol hydrochloride (BIH1526) (Active Comparator): One lozenge 20 mg on as-needed basis, up to 6 times per day
  Interventions: Drug: ambroxol BIH1526
- Placebo (Placebo Comparator): One lozenge on as-needed basis, up to 6 times per day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ambroxol BIH1526 — Pharmaceutical form: lozenges Route of administration: oromucosal
  Arms: Ambroxol hydrochloride (BIH1526)
Drug: placebo — Pharmaceutical form: lozenges Route of administration: oromucosal
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess the efficacy of the new hard boiled Ambroxol lozenges 20 mg for the relief of sore throat pain in patients with acute pharyngitis.

Secondary Objective:

To assess the safety of the new hard boiled Ambroxol lozenges 20 mg in patients with acute pharyngitis.

DETAILED DESCRIPTION:
Duration per participant is up to 4 days.

ELIGIBILITY:
Inclusion criteria:

* Adult male or female patients complaining of sore throat due to acute pharyngitis with an onset no more than 72 hours prior to Visit 1.
* Patients with a score of 6 or greater on a 0-10-point pain intensity numerical rating scale.
* Signed written informed consent.

Exclusion criteria:

Patients suffering from pharyngitis of bacterial origin.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity difference (PID) | hour 3
  Change from baseline to hour 3 in time-weighted average of PID after the first lozenge, expressed as the ratio of the predose baseline, sum of PID (SPIDnorm, 0-3h)

SECONDARY OUTCOMES:
Change in SPID | hour 24
  Change from baseline to hour 24 in time-weighted average of PID after the first lozenge, expressed as the ratio of the predose baseline, sum of PID (SPIDnorm, 0-24h)
3-hour patient assessment of efficacy | hour 3
  Patient assessment of efficacy after 3 hours of the first study drug intake using a 5-point verbal rating scale (VRS) to rate whether the trial medication relieves sore throat pain, where 0 = poor and 4 = excellent
24-hour patient assessment of efficacy | hour 24
  Patient assessment of efficacy after 24 hours of the first study drug intake using a 5-point VRS
Adverse events | baseline to day 4
  Incidence of the adverse events
Patient assessment of tolerability | hour 3, hour 24 and day 2, day 3 or day 4
  Patient assessment of tolerability after 3 hours, Day 1, on Day 2, Day 3 and Day 4 using a 5-point VRS, where 0 = poor and 4 = excellent
Final assessment of tolerability | day 4
  Investigator and patient assessment of tolerability on Day 4 using a 5-point VRS, where 0 = poor and 4 = excellent

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 7100005, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Sousa R, Lakha DR, Brette S, Hitier S. A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Ambroxol Hard-Boiled Lozenges in Patients with Acute Pharyngitis. Pulm Ther. 2019 Dec;5(2):201-211. doi: 10.1007/s41030-019-00100-w. Epub 2019 Oct 18. PMID 32026411